CLINICAL TRIAL: NCT05751070
Title: Comparison of Bowen and Graston Technique in Patients of Tension Neck Syndrome
Brief Title: Bowen and Graston Technique in Patients of Tension Neck Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01396 Amna Jamil
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Neck Syndrome
Keywords: NECK PAIN; NECK DISABILITY; Instrument assisted soft tissue treatment method
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bowen Technique (Active Comparator): BOWEN TECHNIQUE Hot pack TENS Cervical isometrics
  Interventions: Other: Bowen Technique
- Graston technique (Experimental): GRASTON TECHNIQUE Hot pack TENS Cervical isometrics
  Interventions: Other: Graston technique

INTERVENTIONS:
Other: Bowen Technique — They would be receiving conventional treatment as follow:
  Hot pack for 10 minutes TENS for 10 minutes Cervical isometrics 10 reps with 5 sec hold Additionally The Bowen treatment will be 15 to 20 Bowen moves with 2 mins gap between each set for total of 20 mins.
  Arms: Bowen Technique
Other: Graston technique — They would be receiving conventional treatment as follow:
  Hot pack for 10 minutes TENS for 10 minutes Cervical isometrics 10 reps with 5 sec hold Additionally The Graston treatment will be by using lubricant on the skin then a stainless steel instrument to relax the fascia and muscles. The frequency of the plastering and friction movements will be applied in 60 repetitions per minute for total of 20 mins.
  Arms: Graston technique

SUMMARY:
To compare the effects of Bowen and Graston technique in Tension neck syndrome for neck pain , ROM and disability in patients with Tension neck syndrome .

DETAILED DESCRIPTION:
Tension neck syndrome (TNS) is defined as a myofascial pain localized in the neck and shoulder regions. The symptoms include; pain, tenderness, fatigue and stiffness in the neck and shoulder musculature, headaches radiating from the neck, without a history of injury herniated cervical disk, or degenerative processes. It is characterized pain over the neck region and muscle tenderness elicited on palpation and or neck movement. TNS patients with pain have the reduced sensitivity of the neck proprioception. TN may be work- and individual-related and sociopsychological factors may have effect.

Bowen Therapy, is a dynamic fascial and muscle release approach, consisting of gentle cross-fiber movements applied to the fascia, muscles, tendons, muscle insertions, muscle septa, ligaments and viscera.

Grastοn technique is an instrument assisted soft tissue treatment method (ІASTM) derived from the Cyriax1 cross-friction massage. Physіοtherapist strikes stainless steel instrument in a longitudinal dіrectіοn and in circular patterns at the treatment site

ELIGIBILITY:
Inclusion Criteria:

1. Age group 20-45
2. Both males and females
3. Patients diagnosed with VDTS induced Tension neck syndrome in Upper trapezius, SCM & Levator scapulae muscles.
4. Specific criteria will be applied to make diagnosis of Visual display terminal syndrome:

   syndrome, requiring 3 or more symptoms from the following: Patients from Tension neck syndrome such as neck pain, stiffness & tenderness, fatigue or feeling of tiredness, possible headache, pain during movement etc. within past 7 days Musculoskeletal discomfort (pain, tenderness & stiffness)in shoulder, elbow, lower back & wrist/hand regions Ocular symptoms i.e. eye strain or eye dryness from past 7 days
5. Desktop, laptop and excessive smartphone users for more than 2 hours per day at eye level with extreme neck position and static work posture for at least 5 days per week

Exclusion Criteria:

1. Cervical radiculopathy
2. Uncontrolled systemic disease
3. Neck pain due to diabetes, trauma, fracture, infectious or inflammatory process
4. Previous neck or shoulder surgery
5. Patients who are using any medication to reduce the neck pain & discomfort
6. Malignancy

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2023-12-24 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
NPRS FOR NECK PAIN | 2 WEEKS
  The NPRS is a segmented numeric version of the visual analog scale in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.
  The scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")

SECONDARY OUTCOMES:
Range of Motion | 2 WEEKS
  A goniometer is an instrument that measures the available range of motion at a joint.
  Normal range of motion, using the anatomical position as zero degrees.
Neck Disability Index | 2 WEEKS
  Neck Disability Index (NDI) is a questionnaire designed to assess how neck pain has affected patient's ability to manage in everyday life. It has total 10 sections.

CONTACTS AND LOCATIONS:
Overall Officials: KINZA ANWAR, MS-OMPT, Principal Investigator — RIPHAH INTERNATIONAL UNIVERSITY,ISLAMABAD,PAKISTAN
Locations (1):
- WeCare Physiotherapy Clinic, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No